CLINICAL TRIAL: NCT03129022
Title: Failed Epidural Anesthesia During Labor: Evaluation of Risk Factors and Impact on Labor ,Maternal and Fetal Outcomes
Brief Title: Failed Epidural Anesthesia During Labor: Evaluation of Risk Factors and Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 168
Record Dates: First submitted 2017-04-19; First posted 2017-04-26 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Vaginal Delivery
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successful epidural anaesthesia (Active Comparator): It is defined as VAS score <5, 30 min after a loading dose, given after the last attempt.
  Interventions: Procedure: epidural anaesthesia
- Failed epidural anaesthesia (Active Comparator): It is defined as VAS score ≥5, 30 min after a loading dose, given after the last attempt.
  Interventions: Procedure: epidural anaesthesia

INTERVENTIONS:
Procedure: epidural anaesthesia — Women requesting epidural analgesia received a bolus of intravenous infusion of lactated Ringer's solution before initiation of the procedure. An 18-gauge Tuohy needle and closed-tip clear catheter with three lateral orifices were used in the sitting or lateral position, with a loss-of-resistance to air technique. Epidural catheters were routinely inserted 5-6 cm inside the epidural space. A test dose of 2 ml of lidocaine 2% was initiated followed by a loading dose of 10 ml of bupivacaine 0.25%. Analgesia is maintained throughout labor using 0.125% bupivacaine with fentanyl 2 μg/ml with patient-controlled epidural analgesia by means of a continuous epidural infusion (8 ml/h basal rate) and patient-controlled boluses (3 ml each) with 20-minlock-out intervals

SUMMARY:
Women requesting epidural analgesia will receive a bolus of intravenous infusion of lactated Ringer's solution before initiation of the procedure. An 18-gauge Tuohy needle and closed-tip clear catheter with three lateral orifices (Portex, Smith Medical, Hythe, UK) were used in the sitting or lateral position, with a loss-of-resistance to air technique. Epidural catheters will be inserted 5-6 cm inside the epidural space. A test dose of 2 ml of lidocaine 2% iss initiated followed by a loading dose of 10 ml of bupivacaine 0.25%. Analgesia is established and maintained throughout labor and delivery using 0.125% bupivacaine with fentanyl 2 μg/ml with patient-controlled epidural analgesia by means of a continuous epidural infusion (8 ml/h basal rate) and patient-controlled boluses (3 ml each) with 20-minlock-out intervals, continued at the same bolus dose until delivery.

Pain was evaluated using a 0-10 cm visual analogue scale (VAS) before, 15 and 30 min after the loading dose followed by hourly assessment until delivery. VAS score assessment was based specifically on abdominal or back pain resulting from contractions

DETAILED DESCRIPTION:
Women requesting epidural analgesia will receive a bolus of intravenous infusion of lactated Ringer's solution before initiation of the procedure. An 18-gauge Tuohy needle and closed-tip clear catheter with three lateral orifices (Portex, Smith Medical, Hythe, UK) were used in the sitting or lateral position, with a loss-of-resistance to air technique. Epidural catheters will be inserted 5-6 cm inside the epidural space. A test dose of 2 ml of lidocaine 2% iss initiated followed by a loading dose of 10 ml of bupivacaine 0.25%. Analgesia is established and maintained throughout labor and delivery using 0.125% bupivacaine with fentanyl 2 μg/ml with patient-controlled epidural analgesia by means of a continuous epidural infusion (8 ml/h basal rate) and patient-controlled boluses (3 ml each) with 20-minlock-out intervals, continued at the same bolus dose until delivery.

Pain was evaluated using a 0-10 cm visual analogue scale (VAS) before, 15 and 30 min after the loading dose followed by hourly assessment until delivery. VAS score assessment was based specifically on abdominal or back pain resulting from contractions. Failed epidural is defined as VAS score ≥5, 30 min after a loading dose, given after the last attempt. Women who had a repeated attempt due to VAS ≥5 at 30 min or dural puncture or required repositioning of the catheter, resulting in subsequent pain relief expressed as VAS score <5 were not considered to have a Failed epidural. VAS score is assessed by obstetrician and not the anesthesiologist who performed the block. Furthermore, intrapartum vaginal examinations to assess cervical dilatation and fetal head station were also performed by experienced obstetrician.

As part of the study, the women's satisfaction was assessed the morning following delivery using a 1-5 satisfaction scale, where score 1 corresponded to very unsatisfied and score 5 corresponded to very satisfied. Before satisfaction assessment, all women who agreed to participate signed an informed consent and then relevant data was collected from the participants' medical charts.

ELIGIBILITY:
Inclusion Criteria:

* ≥34 weeks of gestation
* receiving epidural analgesia during labor,

Exclusion Criteria:

* Women who had a planned cesarean delivery,
* intrauterine fetal death
* non-vertex presentation
* delivered at less than 30 min after epidural insertion
* contraindication for epidural analgesia (i.e., thrombocytopenia <100,000 cells/μl, ongoing thromboprophylaxis with low-molecular-weight or unfractionated heparin, and bacteremia or infection at the needle-puncture site)

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 500 (Estimated)
Dates: Start 2017-04-30 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
duration of first stage of labor | from start of cervical dilatation till full cervical dilatation
  effect of success and failure of epidural on duration of first stage of labor (..before, 15 and 30 min after the loading dose followed by hourly assessment until delivery..)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Ahmed Maged, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided